CLINICAL TRIAL: NCT07278635
Title: Rewiring the Senses: The Impact of Sensory Integration Therapy on Balance and Cognition in Cerebral Palsy
Brief Title: Sensory Integration Therapy and Function in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sensory process
Record Dates: First submitted 2025-11-17; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy (CP); Balance; Sensory Integration Disorder
Keywords: Cerebral palsy; sensory integration therapy; DOTCA-Ch; balance; functional independence level; sensory processsing
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blind (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Participants in this group will receive individualized sensory integration therapy in addition to standard balance and coordination exercises.
  Therapy will be administered once a week for 45 minutes for a total duration of 12 weeks. Each session will include activities designed to stimulate vestibular, proprioceptive, and tactile systems to improve motor coordination, postural control, sensory processing, and cognitive function.
  Interventions: Behavioral: Sensory Integration Therapy; Behavioral: Balance and Coordination Exercises
- control group (Active Comparator): Participants in this group will receive balance and coordination exercises without sensory integration therapy.
  Exercises will be conducted once a week for 45 minutes over a period of 12 weeks and will include dynamic balance training, postural control activities, and coordination drills appropriate to the participant's functional level.
  Interventions: Behavioral: Balance and Coordination Exercises

INTERVENTIONS:
Behavioral: Sensory Integration Therapy — To evaluate the additional effect of sensory integration therapy on motor, sensory, and cognitive outcomes.
  Arms: Study group
Behavioral: Balance and Coordination Exercises — To assess the effect of standard balance/coordination training without sensory integration.

SUMMARY:
Cerebral palsy (CP) is a non-progressive neurological disorder that affects movement, posture, and functional abilities. Children with CP frequently experience impairments in motor control, sensory processing, balance, postural stability, and cognitive functioning. Sensory integration therapy (SIT) is a therapeutic approach designed to improve the processing and organization of sensory information and may support motor planning and functional performance.

This randomized controlled study aims to examine the effects of sensory integration therapy combined with balance and coordination exercises in children with spastic-type cerebral palsy. Participants will be randomly assigned to receive either balance and coordination training alone or in combination with sensory integration therapy for a 12-week period.

Primary outcomes include balance, functional mobility, and functional independence. Secondary outcomes include sensory processing patterns and cognitive performance. All assessments will be conducted at baseline and following the intervention period by blinded evaluators. The study seeks to provide additional evidence regarding the potential benefits of sensory-based therapeutic approaches within pediatric rehabilitation for children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is characterized by permanent disorders of movement and posture resulting from non-progressive disturbances in the developing fetal or infant brain. Children with CP frequently exhibit motor impairments, sensory processing difficulties, deficits in postural control, and limitations in functional activities. Sensory integration therapy (SIT) is a neurodevelopmental intervention designed to improve the brain's ability to process and organize sensory information, particularly vestibular, proprioceptive, tactile, and visual inputs. Although SIT is commonly used in pediatric rehabilitation, evidence regarding its effects on balance, sensory processing, functional independence, and cognitive skills in children with CP remains limited.

This randomized controlled study aims to evaluate the effects of sensory integration therapy combined with a structured balance and coordination exercise program in children with spastic-type cerebral palsy. Participants will be assigned to either a study group receiving both sensory integration therapy and balance/coordination exercises or a control group receiving only balance/coordination exercises. The intervention will last 12 weeks, with one 45-minute session per week for each component of the program.

Primary outcomes include balance, functional mobility, and functional independence, assessed using the Pediatric Berg Balance Scale (PBBS), the Timed Up and Go Test (TUG), and the Functional Independence Measure for Children (WeeFIM), respectively. Secondary outcomes include sensory processing, evaluated with the Sensory Profile, and cognitive abilities, assessed with the Dynamic Occupational Therapy Cognitive Assessment for Children (DOTCA-Ch). All assessments will be conducted before and after the 12-week intervention period by evaluators blinded to group allocation.

The study is designed to contribute to expanding knowledge on sensory-based rehabilitation strategies and to clarify the potential added value of sensory integration therapy within multidisciplinary treatment approaches for children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy

Age between 6 and 10 years

Gross Motor Function Classification System (GMFCS) Level I or II Ability to understand and follow verbal instructions No severe visual or hearing impairment that interferes with communication Ability to attend and complete the treatment program within the specified duration Enrollment in a special education and rehabilitation center Parental consent obtained for participation in the study

Exclusion Criteria:

* • Receipt of Botulinum toxin-A (BTX-A) treatment within the past 6 months

  * History of hip, knee, or ankle surgery within the past 12 months
  * Presence of severe intellectual disability that prevents active participation
  * Refusal to participate in the study by the child or parent

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2017-11-05 (Actual); Primary Completion 2019-01-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pediatric Berg Balance Scale (PBBS) at 12 Weeks | Baseline (Week 0) and post-intervention (Week 12)
  PBBS (14 items; total 0-56). Higher scores indicate better balance. Primary endpoint is the change score (Week 12 minus Baseline). Assessed by a blinded outcomes assessor.
Change from Baseline in Functional Independence (WeeFIM Total) at 12 Weeks | Baseline and Week 12
  WeeFIM total score (self-care, mobility, cognition domains; standard scoring). Higher scores indicate greater independence. Primary endpoint is the change score. Assessed by a blinded outcomes assessor.
Change from Baseline in Cognitive Function (DOTCA-Ch Total) at 12 Weeks | Baseline and Week 12
  Dynamic Occupational Therapy Cognitive Assessment for Children (DOTCA-Ch) total score; higher scores reflect better cognitive performance. Primary endpoint is the change score. Assessed by a blinded outcomes assessor.

SECONDARY OUTCOMES:
Change from Baseline in Timed Up and Go (TUG) at 12 Weeks | Baseline and Week 12
  TUG measured in seconds; lower times indicate better functional mobility/agility. Endpoint is change score.
Change from Baseline in Sensory Processing (Sensory Profile-Sensory Seeking Subscale) at 12 Weeks | Baseline and Week 12
  Parent-reported Sensory Profile subscale; scoring per instrument manual. Directionality interpreted per manual (improvement defined a priori in analysis plan). Endpoint is change score.
Change from Baseline in Sensory Profile | Baseline and Week 12
  Parent-reported Sensory Profile subscale; scoring per instrument manual. Directionality interpreted per manual (improvement defined a priori in analysis plan). Endpoint is change score.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The plan for sharing individual participant data (IPD) has not yet been determined.

REFERENCES:
- See also: Related Info — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp